CLINICAL TRIAL: NCT01953874
Title: Cardiovascular Improvements With Minute Ventilation-targeted ASV Therapy in Heart Failure (CAT-HF)
Brief Title: Cardiovascular Improvements With MV ASV Therapy in Heart Failure
Acronym: CAT-HF
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: SERVE-HF results showed ASV increased CV mortality in patients with reduced LVEF
Sponsor: ResMed (Industry)
Collaborators: ResMed Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MA-12-12-01
Record Dates: First submitted 2013-09-23; First posted 2013-10-01 (Estimated); Results first posted 2018-02-28 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-01

CONDITIONS: Acute Decompensated Heart Failure; Sleep Disordered Breathing
Keywords: heart failure; congestive heart failure; acute decompensated heart failure; chronic heart failure; left-sided heart failure; heart failure decompensation; sleep apnea; sleep disordered breathing; central sleep apnea; obstructive sleep apnea; cheyne-stokes respiration
MeSH Terms: conditions — Sleep Apnea Syndromes; Heart Failure; Sleep Apnea, Central; Sleep Apnea, Obstructive; Cheyne-Stokes Respiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MV ASV+OMT (Experimental): Minute Ventilation-targeted adaptive servo-ventilation therapy plus optimized medical treatment
  Interventions: Device: MV ASV; Drug: Optimized Medical Treatment
- OMT only (Active Comparator): Optimized Medical Treatment for heart failure in accordance with applicable guidelines (ACCF/AHA Guideline for the Management of Heart Failure and HFSA Heart Failure Guidelines.
  Interventions: Drug: Optimized Medical Treatment

INTERVENTIONS:
Device: MV ASV — Minute ventilation-targeted servo-ventilation therapy.
  Other Names: VPAP Adapt; AutoSet CS
  Arms: MV ASV+OMT
Drug: Optimized Medical Treatment — Beta Blockers, ACE inhibitor or ARB, loop diuretics and/or spironolactone as appropriate, statin if indicated, aspirin and/or warfarin if indicated

SUMMARY:
The aim of the study is to compare the effects of MV targeted ASV in addition to optimized medical therapy versus optimized medical therapy alone at 6 months in patients with acute decompensated HF. The study will also assess changes in functional parameters, biomarkers, quality of life (QOL), and sleep.

DETAILED DESCRIPTION:
This study is a randomized, unblinded, multi-center trial with parallel group design, with subjects randomized to either control (optimized medical therapy for chronic heart failure) or active treatment (optimized medical therapy plus use of MV-targeted ASV) in a 1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

* Patients 21 years or older
* Patients with prior clinical diagnosis of heart failure (HFrEF or HFpEF), or de novo diagnosis of HFpEF indicated by a local BNP≥300 pg/mL or NT pro-BNP≥1200 pg/mL on admission without systolic blood pressure >180 mmHg or atrial fibrillation, or diagnosis of HFrEF indicated by documented evidence of prescribed beta-blockers and ACE-inhibitors or ARBs for at least 4 weeks prior to admission
* Hospital admission for acute decompensated HF as determined by:

  * Dyspnea at rest or with minimal exertion

    * AND At least two of the following signs and symptoms:
  * Orthopnea
  * Pulmonary rales beyond basilar
  * Chest congestion on x-ray
  * BNP≥300pg/mL or NT pro-BNP≥1200pg/mL
  * Pulmonary capillary wedge pressure (PCWP) ≥25mmHg during current hospitalization
* Presented to hospital or clinic at least 24 hours prior to consent
* Patient stable enough to stop oxygen use for duration of polygraphy test or have access to dual lumen cannula for polygraphy test
* Sleep disordered breathing (SDB) documented by polygraphy with an AHI≥15 events/hour
* Patient is able to fully understand study information and sign a consent form

Exclusion Criteria:

* Right-sided heart failure without left-sided heart failure
* Sustained systolic blood pressure <80 mmHg at baseline
* Acute coronary syndrome within 1 months of randomization
* Active myocarditis
* Complex congenital heart disease
* Constrictive pericarditis
* Non-cardiac pulmonary edema
* Clinical evidence of digoxin toxicity
* Need for mechanical hemodynamic support at time of randomization
* Oxygen saturation ≤85% at rest during the day or at start of nocturnal oximetry recording or regular use of oxygen therapy (day or night)
* COPD exacerbation as the primary reason for hospital admission
* Current use (within 4 weeks of study entry) of any PAP-therapy (eg, fixed, bi-level, or APAP)
* Life expectancy < 1 year for diseases unrelated to HF
* Transient ischemic attack (TIA) or Stroke within 3 months prior to randomization
* CABG procedure within 3 months prior to randomization, or planned to occur during study period
* CRT implant within 3 months prior to randomization , or planned to occur during study period
* VAD implant planned to occur during study period
* Heart transplant list Status 1a or 1b
* Status post-transplant or LVAD
* Prescribed inotrope therapy anticipated at discharge
* Chronic Dialysis
* Known amyloidosis, hypertrophic obstructive cardiomyopathy, arteriovenous fistulas
* Primary hemodynamically significant uncorrected valvular heart disease (obstructive or regurgitant) with planned intervention within 6 months of randomization
* Pregnant, or planning to become pregnant
* Cannot tolerate ASV treatment during run-in
* Cannot perform 6MWT at baseline
* Occupation as a commercial driver or pilot and plan to be performing these activities during the study period
* Inability to comply with planned study procedures
* Participation in pharmaceutical or treatment-related clinical study within 1 month of study enrollment

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2013-12; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher O'Connor, MD, Principal Investigator — Duke University
Locations (15):
- United States (14):
  - The Heart Center, Huntsville, Alabama
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - VA Medical Center, Denver, Colorado
  - Mercer University, Macon, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Maryland, Baltimore, Maryland
  - St. Luke's Hospital of Kansas City, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Penn State Hershey, Hershey, Pennsylvania
  - Jefferson Heart Institute, Philadelphia, Pennsylvania
  - Sentara Cardiovascular Research Institute, Norfolk, Virginia
  - University of Washington, Seattle, Washington
- Heart and Diabetes Center - North Rhine-Westphalia (HDZ-NRW), Bad Oeynhausen, Germany

REFERENCES:
- [Derived] Piccini JP, Pokorney SD, Anstrom KJ, Oldenburg O, Punjabi NM, Fiuzat M, Tasissa G, Whellan DJ, Lindenfeld J, Benjafield A, Woehrle H, Blase A, O'Connor CM. Adaptive servo-ventilation reduces atrial fibrillation burden in patients with heart failure and sleep apnea. Heart Rhythm. 2019 Jan;16(1):91-97. doi: 10.1016/j.hrthm.2018.07.027. Epub 2018 Jul 27. PMID 30059750
- [Derived] O'Connor CM, Whellan DJ, Fiuzat M, Punjabi NM, Tasissa G, Anstrom KJ, Benjafield AV, Woehrle H, Blase AB, Lindenfeld J, Oldenburg O. Cardiovascular Outcomes With Minute Ventilation-Targeted Adaptive Servo-Ventilation Therapy in Heart Failure: The CAT-HF Trial. J Am Coll Cardiol. 2017 Mar 28;69(12):1577-1587. doi: 10.1016/j.jacc.2017.01.041. PMID 28335841
- [Derived] Fiuzat M, Oldenberg O, Whellan DJ, Woehrle H, Punjabi NM, Anstrom KJ, Blase AB, Benjafield AV, Lindenfeld J, O'Connor CM. Lessons learned from a clinical trial: Design, rationale, and insights from The Cardiovascular Improvements with Minute Ventilation-targeted Adaptive Sero-Ventilation (ASV) Therapy in Heart Failure (CAT-HF) Study. Contemp Clin Trials. 2016 Mar;47:158-64. doi: 10.1016/j.cct.2016.01.001. Epub 2016 Jan 19. PMID 26806668

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MV ASV+OMT | OMT Only
Started | 65 | 61
Completed | 65 | 61
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MV ASV+OMT | OMT Only | Total
Number analyzed (Participants) | 65 | 61 | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (13.5) | 63.2 (13.4) | 62.1 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 33
  Male | 49 | 44 | 93
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 0 | 4
  Not Hispanic or Latino | 59 | 60 | 119
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 28 | 23 | 51
  White | 35 | 34 | 69
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 48 | 43 | 91
  Germany | 17 | 18 | 35
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 32.3 (9.0) | 31.4 (8.6) | 31.9 (8.8)
New York Heart Association (NYHA) Class [Count of Participants; unit: Participants] — NYHA Class I: Cardiac disease, but not symptoms and no limitation in ordinary physical activity, e.g. shortness of breath when walking, climbing stairs etc.
  NYHA Class II: Mild symptoms (mild shortness of breath and/or angina) and slight limitation during ordinary activity.
  NYHA Class III: Marked limitation in activity due to symptoms, even during less-than-ordinary activity, e.g. walking short distances (20-100m). Comfortable only at rest.
  NYHA Class IV: Severe limitations. Experiences symptoms even while at rest. Mostly bedbound patients.
  Participants
    NYHA Class I | 3 | 3 | 6
    NYHA Class II | 19 | 11 | 30
    NYHA Class III | 32 | 43 | 75
    NYHA Class IV | 9 | 3 | 12
    Not done | 2 | 1 | 3
Left ventricular ejection fraction (LVEF) [Count of Participants; unit: Participants]
  Reduced ejection fraction (</=45%) | 52 | 50 | 102
  Preserved ejection fraction (>45%) | 13 | 11 | 24
Comorbid Conditions [Number; unit: participants]
  Diabetes mellitus | 35 | 34 | 69
  Hypertension | 52 | 56 | 108
  COPD | 12 | 11 | 23
Ischemic HF etiology [Number; unit: participants] | 26 | 18 | 44
Atrial fibrillation [Number; unit: participants] | 26 | 26 | 52
Implanted device [Number; unit: participants]
  Pacemaker | 3 | 6 | 9
  ICD | 26 | 15 | 41
N-terminal pro-brain natriuretic peptide (NT pro-BNP) [Mean (Standard Deviation); unit: pg/mL] | 3468.5 (4231.6) | 6056.4 (8401.9) | 4752.0 (6734.9)
6-minute walk distance [Mean (Standard Deviation); unit: meters] | 221.4 (122.7) | 196.1 (114.6) | 209.2 (119)
Concomitant medications [Number; unit: participants]
  ACE-I or ARB (HFrEF only) | 39 | 38 | 77
  Beta blocker (HFrEF only) | 47 | 46 | 93
  Aldosterone agonist | 33 | 29 | 62
  Loop diuretic | 58 | 53 | 111

OUTCOME MEASURES:

1. Primary Outcome: Global Rank Endpoint
Description: A rank order response based on survival free from CV hospitalization and improvement in functional capacity measured by 6MWD. All participants were first ranked by time to death, then ranked by time to CV hospitalization, and then ranked by percentage change in 6MWD. For time to event measures (time to death and time to hospitalization), the shorter the amount of time, the lower the rank assigned to that participant. For percentage changes in 6MWD, the smaller the percentage change, the lower the rank assigned to that participant. Each component was then combined to create a rank value that ranged between 0 and 100. Overall, higher rank values are associated with better outcomes.
Time Frame: Baseline, 6 months
Measure: Mean (Standard Deviation); unit: Standardized global rank order value
Arm/Group | MV ASV+OMT | OMT Only
Number analyzed (Participants) | 65 | 61
Standardized global rank order value | 50.4 (28.3) | 49.6 (30.0)
Statistical Analysis 1: Comparison: MV ASV+OMT vs OMT Only; The primary endpoint was a composite measure of global rank order response based on survival time, freedom from CV hospitalization, and improvement in functional capacity measured by percent change in 6MWD from baseline to 6 months. The plan was to randomize up to 215 subjects. However, due to safety issues observed in SERVE-HF, randomization was stopped at 126 subjects; Test type: Other — The primary analysis was based on the Wilcoxon-Mann-Whitney test and therefore the power calculation was approximated using the approach of Tang; p = 0.916, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Six-minute Walk Distance
Description: Change in functional parameters as measured by 6-minute walk test (6MWT)
Time Frame: Change from Baseline to 6 months
Population: Reasons 6MWT was not performed:
  In the MV ASV+OMT arm, 5 were discontinued prematurely, 3 participants could not walk, 4 participants were too critically ill, and 2 participants refused.
  In the OMT only arm, 12 were discontinued prematurely, 1 participant could not walk, and 2 participants refused.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | MV ASV+OMT | OMT Only
Number analyzed (Participants) | 51 | 46
meters | 22.6 (131.3) | 61.2 (117.4)

3. Secondary Outcome: NT Pro-BNP
Description: Change in neurohumoral activation as measured by N-terminal pro b-type natriuretic peptide.
Time Frame: Change from Baseline to 6 months
Population: For endpoints that needed a change in measures from baseline to 6 months, if a subject missed one of the measurements, the subject was excluded from the analysis.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | MV ASV+OMT | OMT Only
Number analyzed (Participants) | 41 | 44
pg/mL | 172.7 (3429.1) | -1069.9 (6768.2)

4. Secondary Outcome: Kansas City Cardiomyopathy Questionnaire (KCCQ)
Description: The KCCQ is a 23-item, self-administered instrument that quantifies physical function, symptoms (frequency, severity and recent change), social function, self-efficacy and knowledge, and quality of life. Scores are transformed to a range of 0-100, in which higher scores reflect better health status.
Time Frame: Change from Baseline to 6 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | MV ASV+OMT | OMT Only
Number analyzed (Participants) | 52 | 49
scores on a scale | 20.3 (28.3) | 24.7 (28.0)

5. Secondary Outcome: Biomarkers - Inflammation
Description: Biomarkers of inflammation reported as troponin I ultra-sensitive
Time Frame: Change from Baseline to 6 months
Population: Not all participants had biomarker samples that were able to be analyzed. For endpoints that needed a change in measures from baseline to 6 months, if a subject missed one of the measurements, the subject was excluded from the analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | MV ASV+OMT | OMT Only
Number analyzed (Participants) | 42 | 44
ng/mL | -13.3 (32.1) | -14.1 (41.8)

6. Secondary Outcome: Biomarkers - Cardiovascular
Description: Biomarkers of cardiovascular function reported as hs-CRP
Time Frame: Change from Baseline to 6 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | MV ASV+OMT | OMT Only
Number analyzed (Participants) | 42 | 44
mg/L | 0.03 (0.6) | 0.29 (1.6)

7. Secondary Outcome: Biomarkers - Renal Function
Description: Biomarkers of renal function reported as creatinine
Time Frame: Change from Baseline to 6 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | MV ASV+OMT | OMT Only
Number analyzed (Participants) | 24 | 18
mg/dL | 0.18 (0.66) | 0.08 (0.38)

8. Secondary Outcome: ECHO Parameters - LVEF
Description: Echocardiographic parameters, including LVEF (left ventricular ejection fraction) and LVESVI (left ventricular end-systolic volume index) for patients with HFrEF (heart failure with reduced ejection fraction), and E/e' (ratio between early mitral inflow velocity and mitral annular early diastolic velocity) for patients with HFrEF or HFpEF (heart failure with preserved ejection fraction).
Time Frame: Change from Baseline to 6 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: %EF
Arm/Group | MV ASV+OMT | OMT Only
Number analyzed (Participants) | 41 | 37
%EF | 3.8 (6.3) | 5.0 (9.5)

9. Secondary Outcome: ECHO Parameters - LVESVI
Description: as for outcome 8
Time Frame: Change from Baseline to 6 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mL/m^2
Arm/Group | MV ASV+OMT | OMT Only
Number analyzed (Participants) | 38 | 35
mL/m^2 | -9.0 (21.1) | -8.6 (16.2)

10. Secondary Outcome: ECHO Parameters - E/e' Ratio
Description: Echocardiographic parameters, including LVEF (left ventricular ejection fraction) and LVESVI (left ventricular end-systolic volume index) for patients with HFrEF (heart failure with reduced ejection fraction), and E/e' (ratio between early mitral inflow velocity and mitral annular early diastolic velocity) for patients with HFpEF (heart failure with preserved ejection fraction).
Time Frame: Change from Baseline to 6 months
Population: For endpoints that needed a change in measures from baseline to 6 months, if a subject missed one of the measurements, the subject was excluded from the analysis. HFrEF and HFpEF subjects were separated accordingly.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | MV ASV+OMT | OMT Only
Number analyzed (Participants) | 39 | 39
ratio
  Change in E/e' (HFpEF): number analyzed (Participants) | 8 | 8
  Change in E/e' (HFpEF) | -2.1 (9.0) | -4.6 (6.7)
  Change in E/e' (HFrEF): number analyzed (Participants) | 31 | 31
  Change in E/e' (HFrEF) | -3.2 (9.6) | -2.6 (13.7)

11. Secondary Outcome: Win Ratio
Description: Patients in the new treatment and control groups are formed into matched pairs based on their risk profiles. For each matched pair, the new treatment patient is labeled a 'winner' or a 'loser' depending on who had a CV death first. If that is not known, they are labeled a 'winner' or 'loser' depending on who had a HF hospitalization first. Otherwise they are considered tied. The win ratio is the total number of winners divided by the total numbers of losers.
Time Frame: 6 months
Measure: Number (95% Confidence Interval); unit: Ratio
Groups:
- All Subjects: Minute Ventilation-targeted adaptive servo-ventilation therapy plus optimized medical treatment compared to optimized medical treatment only
  MV ASV: Minute ventilation-targeted servo-ventilation therapy.
  Optimized Medical Treatment: Beta Blockers, ACE inhibitor or ARB, loop diuretics and/or spironolactone as appropriate, statin if indicated, aspirin and/or warfarin if indicated
Arm/Group | All Subjects
Number analyzed (Participants) | 126
Ratio | 0.97 [0.59 to 1.61]

12. Secondary Outcome: Sleep Parameters
Description: Sleep and sleep disordered breathing parameters (AHI, nocturnal hypoxemia)
Time Frame: Change from Baseline to 6 months
Population: Not all subjects in the active arm successfully measured ODI. For endpoints that needed a change in measures from baseline to 6 months, if a subject missed one of the measurements, the subject was excluded from the analysis.
Measure: Mean (Standard Deviation); unit: events per hour
Arm/Group | MV ASV+OMT | OMT Only
Number analyzed (Participants) | 58 | 42
events per hour
  Change in AHI | -33.7 (16.9) | -17.9 (22.3)
  Change in ODI: number analyzed (Participants) | 38 | 42
  Change in ODI | -28.3 (17.5) | -16.3 (20.5)

13. Secondary Outcome: Number of Subjects With HF Hospitalization
Description: Rates of hospitalization or urgent clinic visit for worsening of heart failure and for any reason
Time Frame: 2 days, 1 week, 1, 2, 3, and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | MV ASV+OMT | OMT Only
Number analyzed (Participants) | 65 | 61
Participants | 34 | 27

14. Secondary Outcome: Death
Description: Rate of Cardiovascular and all-cause death
Time Frame: 2 days, 1 week, 1, 2, 3, and 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | MV ASV+OMT | OMT Only
Number analyzed (Participants) | 65 | 61
Participants | 4 | 7

15. Secondary Outcome: Time Dead/Hospitalized
Description: Total days dead or hospitalized at study end
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: number of days
Arm/Group | MV ASV+OMT | OMT Only
Number analyzed (Participants) | 65 | 61
number of days | 23.9 (39.3) | 24.1 (42.8)

16. Secondary Outcome: DASI
Description: The Duke Activity Status Index is a 12-item patient-reported outcome validated for the assessment of functional capacity based on the ability to perform everyday activities. With a total range of 0 to 58.20, a higher score indicates better quality of life.
Time Frame: Change from Baseline to 6 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | MV ASV+OMT | OMT Only
Number analyzed (Participants) | 52 | 49
scores on a scale | 3.7 (13.4) | 5.2 (14.5)

17. Secondary Outcome: EQ-5D-5L Index
Description: The EQ-5D-5L is a standardized self-report questionnaire that is used as a measure of health outcome. The EQ-5D-5L questionnaire is comprised of the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. Responses were indexed using the EQ-5D-5L US value set to scale the 5 dimensions. A score of -0.109 indicates extreme problems for all dimensions and a score of 1.000 indicates no problems for all dimensions. Therefore, a higher score indicates better general health.
Time Frame: Change from Baseline to 6 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | MV ASV+OMT | OMT Only
Number analyzed (Participants) | 51 | 61
scores on a scale | 0.07 (0.23) | 0.03 (0.22)

18. Secondary Outcome: PHQ-9
Description: The PHQ-9 is the nine item depression scale of the Patient Health Questionnaire. The PHQ-9 is a self-administered instrument for screening, diagnosing, monitoring and measuring the severity of depression. The PHQ-9 incorporates DSM-IV depression diagnostic criteria with other leading major depressive symptoms into a brief self-report tool. The tool rates the frequency of the symptoms which factors into the following scoring severity index: 0 - Not at all, 1 - Several Days, 2 - More than Half the Days, 3 - Nearly Every Day. Total score can range from 0 to 27. A higher score indicates increased severity.
Time Frame: Change from Baseline to 6 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | MV ASV+OMT | OMT Only
Number analyzed (Participants) | 52 | 49
scores on a scale | -2.8 (6.7) | -4.6 (6.7)

19. Secondary Outcome: PSQI
Description: The Pittsburgh Sleep Quality Index is a 19-item subjective measurement of sleep. It is an effective instrument used to measure the quality and patterns of sleep in the older adult. It differentiates "poor" from "good" sleep by measuring seven areas: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication and daytime dysfunction over the last month. The subject self-rates each of these seven areas of sleep. The seven component scores are then added to yield a total score with a range of 0-21 points, "0" indicating no difficulty and "21" indicating severe difficulties in all areas.
Time Frame: Change from Baseline to 6 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | MV ASV+OMT | OMT Only
Number analyzed (Participants) | 48 | 48
scores on a scale | -2.7 (5.0) | -3.3 (4.9)

20. Secondary Outcome: ESS
Description: The Epworth Sleepiness Scale is a simple, 8-item self-administered questionnaire which provides a measurement of the subject's general level of daytime sleepiness. The individual is asked on a scale of 0-3 to score the likelihood of falling asleep in eight various situations. With a total range of 0 to 24, a higher score indicates increased severity.
Time Frame: Change from Baseline to 6 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | MV ASV+OMT | OMT Only
Number analyzed (Participants) | 51 | 48
scores on a scale | -1.6 (5.6) | -2.1 (5.1)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | MV ASV+OMT | OMT Only
All-Cause Mortality (participants affected / at risk) | 4/65 | 7/61
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/61
Other Adverse Events (participants affected / at risk) | 2/58 | 1/61
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MV ASV+OMT (N=58) | OMT Only (N=61)
Bloating (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Weight gain (Cardiac disorders) | 0 (0) | 1 (1)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The trial was terminated early because of the unexpected safety signal reported in SERVE-HF.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No